CLINICAL TRIAL: NCT03412799
Title: Phase 1A/1B Dose Escalation and Expansion Study of SBP-101 in Combination With Nab-Paclitaxel and Gemcitabine in Subjects With Previously Untreated Metastatic Pancreatic Ductal Adenocarcinoma
Brief Title: Study of SBP-101 Combined With Nab-Paclitaxel and Gemcitabine in Pancreatic Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Panbela Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CL-SBP-101-03
Record Dates: First submitted 2018-01-19; First posted 2018-01-26 (Actual); Last update posted 2022-05-25 (Actual); Status verified 2022-05

CONDITIONS: Pancreatic Cancer Metastatic; Pancreatic Cancer Stage IV; Stage IV Pancreatic Cancer
MeSH Terms: conditions — Pancreatic Neoplasms | interventions — 130-nm albumin-bound paclitaxel; Albumin-Bound Paclitaxel; Gemcitabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

INTERVENTIONS:
Drug: SBP-101 — Administered as subcutaneous (SC) injection, escalating dose cohorts
  Other Names: diethyl dihydroxyhomospermine; [(HO)2-DEHSPM]
Drug: nab-paclitaxel — Administered as intravenous (IV) infusion
  Other Names: abraxane; protein-bound paclitaxel
Drug: Gemcitabine Injection — Administered as intravenous (IV) infusion
  Other Names: gemcitabine hydrochloride; Gemzar

SUMMARY:
This is an open-label phase 1A/1B study to assess the safety, tolerability and pharmacokinetics of SBP-101 when combined with nab-paclitaxel and gemcitabine in subjects with previously untreated metastatic pancreatic ductal adenocarcinoma and to identify a recommended phase 2 dose. The study will also assess preliminary efficacy of the 3-drug treatment combination.

DETAILED DESCRIPTION:
The study will be conducted in two phases: dose escalation and expansion. Up to three dose levels of SBP-101 will be assessed in up to 18 subjects during dose escalation. The expansion phase of the study will consist of 10 additional subjects who will receive the recommended dose of SBP-101 combined with nab-paclitaxel and gemcitabine.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically confirmed metastatic pancreatic ductal adenocarcinoma. Patients with pancreatic acinar cell carcinoma may also be included.
* Is previously untreated for metastatic pancreatic ductal adenocarcinoma, was diagnosed within the past 3 months, and is expected to receive standard treatment with gemcitabine and nab-paclitaxel.
* Measurable disease on CT or MRI scan by RECIST v 1.1 criteria.
* ECOG Performance Status 0 or 1.
* Adult, age ≥ 18 years, male or female.
* Females of child-bearing potential must have a negative serum pregnancy test within 14 days prior to start of study treatment and must use an adequate method of contraception during the study. All sexually active males must also use an adequate method of contraception during the study. Female subjects will be considered to be of childbearing potential unless they are postmenopausal (at least 12 months of consecutive amenorrhea, without other known or suspected cause) and over 55 years old or have been sterilized surgically (i.e., bilateral tubal ligation, hysterectomy or bilateral oophorectomy, all with surgery at least one month before dosing).
* Adequate bone marrow, hepatic, renal and coagulation function as defined by the following:

  1. Absolute neutrophil count ≥1.5 x 109/L
  2. Hemoglobin ≥9.0 g/dL (90 g/L)
  3. Platelets ≥100 x 109/L
  4. Aspartate aminotransferase (AST) and alanine aminotransferase (ALT) ≤2.5 x upper limit of normal (ULN) (if no hepatic metastases). If hepatic tumor involvement, AST and ALT ≤5 x ULN.
  5. Bilirubin ≤1.5 x ULN
  6. Prothrombin time (PT) / international normalized ratio (INR) ≤1.5 x ULN if not on anti-coagulants
  7. Calculated creatinine clearance >50 mL/min using the Cockcroft and Gault equation
* QTc interval ≤ 470 msec at Baseline.
* Life expectancy ≥ 3 months.
* Willing and able to provide written informed consent: voluntary agreement to participate in the study following disclosure of risks and procedures required, including possibility of onset of exocrine pancreatic insufficiency with subsequent requirement for life-long pancreatic enzyme replacement.

Exclusion Criteria:

* Evidence of severe or uncontrolled systemic disease or any concurrent condition that, in the opinion of the Investigator or Medical Monitor, makes it undesirable for the subject to participate in the study or that would jeopardize compliance with the protocol. Subjects with pre-existing well-controlled diabetes are not excluded.
* Medical or psychiatric conditions that compromise the subject's ability to give informed consent or to complete the protocol or a history of non-compliance
* Presence of islet-cell or pancreatic neuroendocrine tumor or mixed adenocarcinoma-neuroendocrine carcinoma
* Have symptomatic central nervous system (CNS) malignancy or metastasis. Screening of asymptomatic subjects without history of CNS metastases is not required.
* Serum albumin <30 g/L (3.0 g/dL)
* Evidence of deep vein thrombosis or pulmonary embolism or other thromboembolic event during screening
* Presence of known active bacterial, fungal, or viral infection requiring systemic therapy
* Known active infection with human immunodeficiency virus (HIV), hepatitis B or C
* Presence of interstitial lung disease, pulmonary fibrosis, or pulmonary hypersensitivity reaction
* Myocardial infarction within the last 12 months, severe/unstable angina, symptomatic congestive heart failure New York Heart Association (NYHA) class III or IV
* Maldigestion/malabsorption syndrome pre-dating the diagnosis of pancreatic cancer.
* Pregnant or lactating
* Major surgery within 4 weeks of the start of study treatment, without complete recovery
* Known hypersensitivity to any component of study treatments
* Participation in any other clinical investigation within 4 weeks of receiving the first dose of study drug
* Subjects taking metformin. Diabetics on treatment with metformin, or any other derivative thereof, must discontinue it while on study. (Other diabetic medications are allowed.)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2018-06-04 (Actual); Primary Completion 2022-02-28 (Actual); Study Completion 2022-02-28 (Actual)

PRIMARY OUTCOMES:
Recommended dose of SBP-101 | Up to 12 months following the first dose of treatment

SECONDARY OUTCOMES:
Number of subjects with adverse events as a measure of safety and tolerability | Up to 24 months following the first dose of treatment
Tumor response will be evaluated on RECIST definitions | Every 8 weeks during treatment assessed up to 24 months
Area under the plasma concentration versus time curve (AUC) for all three drugs | Day 1 of Cycle 1
Peak plasma concentration (Cmax) for all three drugs | Day 1 of Cycle 1

CONTACTS AND LOCATIONS:
Overall Officials: Suzanne Gagnon, MD, Study Director — Panbela Therapeutics, Inc.
Locations (7):
- United States (3):
  - Scripps MD Anderson Cancer Center, La Jolla, California
  - University of Florida, Gainesville, Florida
  - University of Rochester Medical Center, Rochester, New York
- Australia (4):
  - Blacktown Cancer & Haematology Centre, Blacktown, New South Wales
  - John Flynn Private Hospital, Tugun, Queensland
  - Ashford Cancer Centre, Kurralta Park, South Australia
  - Austin Health, Heidelberg, Victoria